CLINICAL TRIAL: NCT02520895
Title: Immunological Repertoire in Patients With Lymphoma and Chronic Lymphocytic Leukemia, Biomedical Research on Medical Devices Human ImmunTracker and Human Immun'IgH
Brief Title: Immunological Repertoire in Patients With Lymphoma and Chronic Lymphocytic Leukemia
Acronym: RIPAL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2009.548; 2010-A00591-38 (Other: ANSM)
Record Dates: First submitted 2014-09-15; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: LYMPHOMA
Keywords: Chronic Lymphocytic Leukemia; Non-Hodgkin lymphoma; Follicular Lymphoma; Diffuse Large B Cell Lymphoma; MALT Lymphoma; T Cell Lymphoma; Immune Repertoire; Infection; relapse; survival; treatment response; VJ rearrangement
MeSH Terms: conditions — Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell; Infections; Recurrence | interventions — Cordocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- large B lymphoma cells (group 1): 30 patients with large B lymphoma cells at diagnosis and who will receive an immunochemotherapy treatment patients will have blood samplings
  Interventions: Biological: blood samplings
- indolent B-cell lymphomas (group 2): 30 patients with indolent B-cell lymphomas without invasion excess blood lymphoma 1 giga / L at diagnosis and who will receive an immunochemotherapy treatment- patients will have blood samplings
  Interventions: Biological: blood samplings
- indolent B-cell lymphomas (group 3): 20 Patients with indolent B-cell lymphomas with lymphocytosis (> 1 Giga / L) at diagnosis and who will receive an immunochemotherapy treatment- patients will have blood samplings
  Interventions: Biological: blood samplings
- Lymphocytic Leukemia Chronic (LLC) (group 4): 20 patients with LLC never treated before and will receive an immunochemotherapy treatment (fludarabine +/- endoxan +/- rituximab or alemtuzumab)- patients will have blood samplings
  Interventions: Biological: blood samplings
- T-cell lymphoma (group 5): 10 Patients with T-cell lymphoma in 1st line therapy and will receive a combination of chemotherapy- patients will have blood samplings
  Interventions: Biological: blood samplings
- follicular lymphoma (group 6): 6 patients with follicular lymphoma in first line or relapsed and will receive a single immunotherapy treatment (rituximab)- patients will have blood samplings
  Interventions: Biological: blood samplings
- Lymphocytic Leukemia Chronic (LLC) (group 7): 6 patients with LLC never treated and will receive a combination of rituximab, fludarabine, endoxan- patients will have blood samplings
  Interventions: Biological: blood samplings
- Lymphocytic Leukemia Chronic (LLC) (group 8): 6 patients with LLC stage A followed for a period of 18 months without treatment- patients will have blood samplings
  Interventions: Biological: blood samplings

INTERVENTIONS:
Biological: blood samplings — patients will have blood samplings at different time : D0: day of inclusion = day of the first course of chemotherapy or the 1st day of the confirmation of the diagnosis (group 8) M3: 3 months (+/- 1 month) after the start of treatment (except for group 8) M6: 6 months (+/- 1 month) after the start of treatment or after the 1st day of the confirmation of the diagnosis (group 8) M12 : 12 months after the start of treatment (group 6 and 7) M18: 18 months (+/- 1 month) after the start of treatment or after the 1st day of the confirmation of the diagnosis (group 8) R: to relapse if it occurs before 18 months or at the time of first treatment if it occurs before 18 months (group 8)

SUMMARY:
RIPAL is a prospective cohort study, which main goal is to define T and B immune repertoire diversity and magnitude in patients with non-Hodgkin lymphoma of high and low grade and chronic lymphocytic leukemia before and after treatment, and to evaluate the association of these parameters with clinical patient data and outcomes.

DETAILED DESCRIPTION:
Constitution of a prospective cohort of 128 patients with 8 different groups of patients. This protocol is designed to evaluate a new tool for detecting the diversity of the repertoire T and B in patients with hematological disease. This in vitro diagnostic device is consisting of molecular biology kits Human ImmunTraCkeR® and Human Immun'IgH® and the analysis tool NDL®

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Subjects with a diagnosis of large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma, MALT, marginal zone, Waldenstrom's disease, chronic lymphocytic leukemia, T-cell lymphoma, anaplastic, cytotoxic or peripheral unspecified angioimmunoblastic.
* Have signed an informed consent for participation in the study and preservation of blood samples for biomedical research.
* Accept to appear in consultation biological samples at the sampling points corresponding to its group.
* The benefits of social security.

Exclusion Criteria:

* Subjects with a diagnosis of Hodgkin disease
* Subjects with a diagnosis of T-prolymphocytic leukemia
* Subjects with a diagnosis of Burkitt's lymphoma
* Subjects with a diagnosis of lymphoblastic lymphoma
* Subjects who had prior-treatment for hematological disease
* Patients under judicial safeguards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with lymphoma or chronic lymphocytic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
change in variations of the T and B cell repertoire in patients with lymphoid blood disease under treatment | from D0 to 18 months
  results given by the technical Immun'IgH® Human and Human ImmunTraCkeR® and score NDL®
  The 2 criteria for obtaining the data are the diversity and intensity of the immune repertoire:
  The intensity of the signal corresponds to the frequency of VJ rearrangements detected in the samples. It is expressed in Arbitrary Units.
  The diversity corresponds to the number of different VJ rearrangements detected compared to all theoretical VJ rearrangement. It is expressed in percentage.

SECONDARY OUTCOMES:
performance of the mapping of the immune repertoire to predict treatment response | from D0 to 18 months
  The response to initial treatment will be confronted with the results given by the technical Immun'IgH® Human and Human ImmunTraCkeR® and score NDL®
  Response to treatment will be assessed by the local treating physician as complete response (CR), unconfirmed complete response (CRu), partial response (PR), stable disease, or progressive disease (PD) in accordance with the International Workshop Standardized Response Criteria for Non-Hodgkin Lymphoma and International Workshop Standardized Response Criteria for Chronic Lymphocytic Leukemia.
performance of the mapping of the immune repertoire to predict progression free survival | from D0 to progression
  the progression free survival will be confronted with the results given by the technical Immun'IgH® Human and Human ImmunTraCkeR® and score NDL®
  For all groups except group 8 (LLC untreated): the progression free survival is defined as the number of months elapsed between the first day of treatment (D0) and progression For The group 8: the progression free survival is defined as the number of months elapsed between the first day of the consultation (D0) that led to the confirmation of diagnosis and the date of first treatment.
performance of the mapping of the immune repertoire to predict the risk of infection | from D0 to 18 months
  the number of patients with infection will be confronted with the results given by the technical Immun'IgH® Human and Human ImmunTraCkeR® and score NDL® All presumed or confirmed infections such as isolated febrile events associated or not with an identifiable site of infection and/or germ clearly identified
sensitivity of detection of the circulating clones | from D0 to 18 months
  results given by the technical Immun'IgH® Human and Human ImmunTraCkeR® and score NDL® will be compared with data obtained from conventional immunophenotypic and molecular data.
  The 3 conventional technics are : morphological examination, immunophenotyping, molecular biology by BIOMED2 primers

CONTACTS AND LOCATIONS:
Overall Officials: Gilles SALLES, MD, Principal Investigator — Service d'Hématologie Clinique, Centre Hospitalier Lyon Sud, France
Locations (1):
- Service d'Hématologie Clinique, Centre Hospitalier Lyon Sud, Pierre-Bénite, France